CLINICAL TRIAL: NCT05413018
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Compare Efficacy and Safety of Oral Azacitidine (CC-486) Plus Best Supportive Care Versus Best Supportive Care as Maintenance Therapy in Chinese Patients With Acute Myeloid Leukemia in Complete Remission
Brief Title: An Efficacy and Safety Study of Oral Azacitidine (CC-486) as Maintenance Therapy in Chinese Participants With Acute Myeloid Leukemia in Complete Remission
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA055-006
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Azacitidine; CC-486; Onureg; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cc-486; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CC-486/Oral Azacitidine Administration (Experimental)
  Interventions: Drug: CC-486
- Placebo Administration (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-486 — Specified dose on specified days
  Other Names: Azacitidine; Onureg
  Arms: CC-486/Oral Azacitidine Administration
Other: Placebo — Specified dose on specified days
  Arms: Placebo Administration

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Oral Azacitidine (CC-486) in Chinese participants with acute myeloid leukemia in complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically confirmed de novo acute myeloid leukemia (AML) or AML secondary to prior myelodysplastic disease or chronic myelomonocytic leukemia (CMML)
* Eastern cooperative oncology group performance status of 0, 1, or 2
* Has undergone induction therapy with intensive chemotherapy with or without consolidation therapy
* Must have achieved first complete remission (CR) or complete remission with incomplete blood count recovery (CRi) status within 6 months (+/- 7 days) prior to starting study therapy

Exclusion Criteria:

* Suspected or proven acute promyelocytic leukemia or acute myeloid leukemia with previous hematologic disorder such as chronic myeloid leukemia or myeloproliferative neoplasms, excluding myelodysplastic syndromes and chronic myelomonocytic leukemia
* Candidate for allogeneic bone marrow or stem cell transplant at screening
* Have achieved CR/CRi following therapy with hypomethylating agents
* AML associated with inv(16), t(8;21), t(16;16), t(15;17), or t(9;22) karyotypes or molecular evidence of such translocations
* Proven central nervous system leukemia
* Prior bone marrow or stem cell transplantation

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | Up to 30 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 42 months
Time to relapse | Up to approximately 30 months
Time to discontinuation of treatment | Up to approximately 42 months
Number of participants with adverse events (AEs) | Up to approximately 42 months
Number of participants with physical examination abnormalities | Up to approximately 42 months
Number of participants with vital sign abnormalities | Up to approximately 42 months
Number of participants with clinical laboratory abnormalities | Up to approximately 42 months
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-t)) | Up to 8 weeks
Maximum observed plasma concentration (Cmax) | Up to 8 weeks
Time of maximum observed concentration (Tmax) | Up to 8 weeks
Terminal elimination half-life (T1/2) | Up to 8 weeks
Minimal/measurable residual disease (MRD) assessment by flow cytometric analysis of hematopoietic cell immunophenotypes | Up to approximately 30 months
Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale | Up to approximately 30 months
EQ-5D-5L scale | Up to approximately 30 months
Visual analog scale (VAS) | Up to approximately 30 months
Healthcare Resource Utilization (HRU): Rate of Hospital Events Per Year | Up to approximately 30 months
  HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the participant. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.
Healthcare Resource Utilization (HRU): Number of Medications | Up to approximately 30 months
  HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the participant. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.
Healthcare Resource Utilization (HRU): Rate of Clinic Visits Per Year | Up to approximately 30 months
  HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the participant. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.
Healthcare Resource Utilization (HRU): Rate of Medical/Diagnostic Events Per Year | Up to approximately 30 months
  HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the participant. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.
Healthcare Resource Utilization (HRU): Number of Treatments for AEs Per Year | Up to approximately 30 months
  HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the participant. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- China (34):
  - Local Institution - 0031, Hefei, Anhui
  - Local Institution - 0013, Beijing, BJ
  - Local Institution - 0027, Beijing, BJ
  - Local Institution - 0028, Chongqing, CQ
  - Local Institution - 0003, Guangzhou, GD
  - Local Institution - 0008, Guangzhou, GD
  - Local Institution - 0010, Shenzhen, GD
  - Local Institution - 0002, Shijiazhuang, HE
  - Local Institution - 0022, Xuzhou, Jiangsu
  - Local Institution - 0005, Shenyang, Liaoning
  - Local Institution - 0020, Shenyang, LN
  - Local Institution - 0016, Chengdu, SC
  - Local Institution - 0006, Shanghai, SH
  - Local Institution - 0030, Xi'an, SN
  - Local Institution - 0033, Taiyuan, SX
  - Local Institution - 0001, Tianjin, TJ
  - Local Institution - 0009, Ürümqi, Xinjiang
  - Local Institution - 0007, Wenzhou, ZJ
  - Local Institution - 0017, Changchun
  - Local Institution - 0019, Changsha
  - Local Institution - 0015, Changsha
  - Local Institution - 0035, Ganzhou
  - Local Institution - 0012, Guangzhou
  - Local Institution - 0014, Hangzhou
  - Local Institution - 0032, Harbin
  - Local Institution - 0011, Jinan
  - Local Institution - 0024, Kunming
  - Local Institution - 0026, Lanzhou
  - Local Institution - 0018, Nanchang
  - Local Institution - 0029, Nanjing
  - Local Institution - 0021, Suzhou
  - Local Institution - 0023, Tianjin
  - Local Institution - 0034, Zhangzhou
  - Local Institution - 0004, Zhengzhou

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html